CLINICAL TRIAL: NCT04777019
Title: Computer Aided Polyp Detection (C3PO) Trial: A Multicenter International Trial Evaluating Diagnostic Accuracy of Artificial Intelligence System in Detecting Colon Polyps
Brief Title: Computer Aided Polyp Detection (C3PO) Trial
Status: Withdrawn | Type: Observational
Why Stopped: Study device not available
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nirav C Thosani, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-20-0687
Record Dates: First submitted 2021-02-02; First posted 2021-03-02 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable as standard of care Colonoscopy — Not applicable since not an intervention

SUMMARY:
Computer aided detection (CADe) algorithms have been developed to overcome human errors and assist endoscopists in detecting more polyps during colonoscopy. The aim of this study was to investigate the accuracy of the novel Pentax Discovery CADe system (Discovery-AI) against pre-recorded videos of colon polyps of various size, shape and pathology while using videos of normal colon segments as controls from two different institutes.

DETAILED DESCRIPTION:
Details regarding polyp size and location, morphology including Paris classification, optical assessment, and bowel preparation were prospectively collected and recorded in the online Redcap software. Final results of polyp histology were also collected. The video library was then independently reviewed for quality assessment by 3 experienced gastroenterologists. Videos that passed the initial quality assessment were then independently evaluated using the Discovery-AI system.

Aim of the study was to evaluate overall performance of Discovery-AI system for polyps of various size, morphology and pathology utilizing a prospectively developed video library.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for a regular or screening colonoscopy at the institution as standard of care.
* Over 18 years of age

Exclusion Criteria:

* None if they qualify based on inclusion criteria
* Pregnant patients
* Inmate or prisoners
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Currently, the most commonly used quality marker in conventional colonoscopy (CC) is adenoma detection rate (ADR), which has been shown to inversely correlate with the incidence of CRC.3 Although colonoscopy is generally considered to be the most accurate screening modality, a substantial number of polyps are still missed. Hence population scheduled for a colonoscopy at either of the institution were part of the project.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-06-07 (Actual); Primary Completion 2023-06-07 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
To investigate the accuracy of the novel Pentax Discovery CADe system (Discovery-AI) against pre-recorded videos of colon polyps of various size, shape and pathology while using videos of normal colon segments as controls | 3 years
  The video library was developed during screening and surveillance colonoscopy and included details on polyp size, location, morphology, overall Boston bowel preparation score (BBPS) and segmental BBPS. Each video segments ranged from 35 seconds to 75 seconds. Before inclusion, each video was evaluated by 3 expert endoscopists individually to assess overall quality of the video. Quality of video was assessed based on pixel resolution and aspect ratio, bowel preparation, overall speed of withdrawal, colon distension, and adequate mucosal exposure. If the video was deemed of adequate quality by at least 2 endoscopists, it was included in the study cohort.

IPD SHARING:
Plan to Share IPD: Undecided